CLINICAL TRIAL: NCT05070598
Title: A Prospective, Single-arm, Phase II Study of Camrelizumab Combined With Pyrotinib Maleate, Nab-paclitaxel and Tegafur Chemotherapy in First-line Treatment of HER2-positive Gastric Cancer
Brief Title: Camrelizumab Combined With Chemotherapy in First-line Treatment of HER2-positive Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Chief Physician, Shengjing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shengjing-LCG
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: HER2-positive Gastric Cancer
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Tegafur

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab +Pyrotinib + Nab-paclitaxel + Tegafur (Experimental): Camrelizumab Q3W d1 Pyrotinib d1-21 Nab-paclitaxel Q3W d1 Tegafur d1-14
  Interventions: Drug: Camrelizumab +Pyrotinib + Nab-paclitaxel + Tegafur

INTERVENTIONS:
Drug: Camrelizumab +Pyrotinib + Nab-paclitaxel + Tegafur — Camrelizumab was given in the first day of each cycle,Nab-paclitaxel was given in the first day of each cycle, Pyrotinib was given everyday of each cycle, Tegafur given in the day 1-14 of each cycle

SUMMARY:
According to the investigator's judgment, there are concomitant diseases that seriously endanger the patient's safety, or affect the patient's completion of the study (such as uncontrolled hypertension, diabetes, thyroid disease, etc.);

ELIGIBILITY:
Inclusion Criteria:

- rious hepatic and renal impairment, organ function must meet the following requirements: ANC ≥ 1.5 × 109/L; PLT ≥ 90 × 109/L; Hb ≥ 90g/L; TBIL ≤ 1.5 × ULN; ALT and AST ≤1.5 × ULN, ALP ≤ 2.5 × ULN; for patients with liver metastases, ALT and AST ≤ 5 × ULN BUN and Cr ≤ 1 × ULN and cre

Exclusion Criteria:

* rious hepatic and renal impairment, organ function must meet the following requirements: ANC ≥ 1.5 × 109/L; PLT ≥ 90 × 109/L; Hb ≥ 90g/L; TBIL ≤ 1.5 × ULN; ALT and AST ≤1.5 × ULN, ALP ≤ 2.5 × ULN; for patients with liver metastases, ALT and AST ≤ 5 × ULN BUN and Cr ≤ 1 × ULN and cre

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
ORR (Objective control rate) | up to 12 months
  The rate of CR and PR, determined using RECIST v1.1 criteria

SECONDARY OUTCOMES:
DCR (Disease control rate) | up to 12 months
  The rate of CR, PR plus SD
PFS (Progression-Free survival) | up to 12 months
  From the date Into this study (signed ICF) to tumor progression or death for any
OS(Overall survival) | up to approximately 24 months
  Baseline until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Caigang Liu, doctor, Study Chair — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, China